CLINICAL TRIAL: NCT04082039
Title: The Efficacy of New Design Dual Channel Elastomeric Pump for Intravenous Patient-controlled Analgesia After Total Laparoscopic Hysterectomy: a Randomized, Double-blind, Prospective Study
Brief Title: Two-channel Intravenous Patient-controlled Analgesia (IV-PCA) After Total Laparoscopic Hysterectomy (TLH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Seok Kyeong Oh, Clinical Assistant Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2019GR0294
Record Dates: First submitted 2019-09-04; First posted 2019-09-09 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Total Laparoscopic Hysterectomy; Patient-controlled Analgesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1-channel PCA (Active Comparator): Ch-1: fentanyl 16 µg/kg, ketorolac 2 mg/kg, ondansetron 12 mg (total volume 100 ml with normal saline) Ch-2: 100ml normal saline only (for blinding)
  Interventions: Other: convetional PCA method unsing only 1-channel
- 2-channel PCA (Experimental): Ch-1: fentanyl 16 µg/kg (total volume 100 ml with normal saline) Ch-2: ketorolac 2 mg/kg, ondansetron 12 mg (total volume 100 ml with normal saline)
  Interventions: Other: utilizing 2-channel

INTERVENTIONS:
Other: convetional PCA method unsing only 1-channel — Ch-1 (flow 2 ml/hr with bolus 2ml/30min lock-out): fentanyl 16 µg/kg, ketorolac 2 mg/kg, ondansetron 12 mg (total volume 100 ml with normal saline); Ch-2 (flow 2ml/h): 100ml normal saline only (for blinding)
  Arms: 1-channel PCA
Other: utilizing 2-channel — Ch-1 (flow 2 ml/hr with bolus 2ml/30min lock-out): fentanyl 16 µg/kg (total volume 100 ml with normal saline; Ch-2 (flow 2ml/h fixed): ketorolac 2 mg/kg, ondansetron 12 mg (total volume 100 ml with normal saline)
  Arms: 2-channel PCA

SUMMARY:
The purpose of this study is to compare the dual channel intravenous patient-controlled analgesia (IV-PCA) with single channel elastomeric pump (only one channel of dual channel pump is used for blinding and the other channel is filled with same volume of saline) in patients undergoing total laparoscopic hysterectomy, in terms of quality of recovery, efficacy of postoperative pain, drug consumption, adverse event, and patient subjective satisfaction.

DETAILED DESCRIPTION:
The Bellomic® M silicone balloon infuser, dual continuous petite type (cebika, Uiwang-si, Gyeonggi-do, Republic of Korea) is a newly designed IV-PCA device that is a 2-channel infusion elastomeric pump with two balloon chambers.

Conventional elastomeric IV-PCA devices were administered with a mixture of drugs in one chamber; when severe opioid related side effects occur, the IV-PCA administration is suspended by clipping, in this situation, not only the analgesic effect of opioid but also the effect of adjuvants could not be applied.

On the other hand, this newly designed device can be controlled as needed by administering adjuvant analgesics or antiemetic agents through another adjustable chamber. It will be expected that facilitate the pain management and increased the patient satisfaction and recovery.

ELIGIBILITY:
Inclusion Criteria:

* patient who was scheduled to undergo elective TLH under general anesthesia, was a female aged 19-75 years, and had an American Society of Anesthesiologists physical status I-II

Exclusion Criteria:

* body mass index > 30.0 kg/m2, known hypersensitivity to the drugs used in this study, significant liver or renal dysfunction, or a history of drug abuse or dependence, recent major procedure or surgery, or preoperative analgesic use

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Korean version of the Quality of Recovery-40 questionnaire (QoR-40K) score | At postoperative 24 hour
  Patient recovery measured by QoR-40K score (maximum score 200)

SECONDARY OUTCOMES:
Pain level was evaluated according to a numeric rating scale | At 6, 12, 24, 36, 48 hours after surgery
  (NRS; 0-100; no pain [0] to worst pain imaginable [100])
Cumulative consumption of PCA over 48 hours | At postoperative 48 hour
The patient's overall satisfaction score | At postoperative 48 hour
  (0-10; 0 = un-satisfied to 10 = full-satisfied)
Occurrence of adverse effects | Participants will be followed for their entire hospital stay, an expected average of 3-4 days
  nausea and vomiting, dry mouth, dizziness, urinary retention, headache, sedation, itchiness, shivering, respiratory depression, confusion, hypotension, and bradycardia

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
In order to protect patient priavacy and personal information, we will limit the provision of individual participant data

REFERENCES:
- [Derived] Oh SK, Kim H, Kim YS, Lee CH, Oh JS, Kwon DH. The effect of newly designed dual-channel elastomeric pump for intravenous patient-controlled analgesia after total laparoscopic hysterectomy: a randomized, double-blind, prospective study. Perioper Med (Lond). 2022 Oct 12;11(1):52. doi: 10.1186/s13741-022-00282-z. PMID 36224646